CLINICAL TRIAL: NCT03017820
Title: Phase I Trial of Systemic Administration of Vesicular Stomatitis Virus Genetically Engineered to Express NIS and Human Interferon, in Patients With Relapsed or Refractory Multiple Myeloma, Acute Myeloid Leukemia, Lymphomas, or Histiocytic/Dendritic Cell Neoplasms
Brief Title: A Vaccine (VSV-hIFNβ-NIS) With or Without Cyclophosphamide and Combinations of Ipilimumab, Nivolumab, and Cemiplimab in Treating Relapsed or Refractory Multiple Myeloma, Acute Myeloid Leukemia or Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1684; R01CA262613 (NIH); P50CA186781 (NIH); NCI-2017-00049 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1684 (Other: Mayo Clinic); 16-005474 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: B-Cell Non-Hodgkin Lymphoma; Histiocytic and Dendritic Cell Neoplasm; Myelodysplastic Syndrome; Previously Treated Myelodysplastic Syndrome; Recurrent Adult Acute Myeloid Leukemia; Recurrent Anaplastic Large Cell Lymphoma; Recurrent Angioimmunoblastic T-Cell Lymphoma; Recurrent Mycosis Fungoides; Recurrent Plasma Cell Myeloma; Recurrent Primary Cutaneous T-Cell Non-Hodgkin Lymphoma; Recurrent T-Cell Non-Hodgkin Lymphoma; Refractory Acute Myeloid Leukemia; Refractory Anaplastic Large Cell Lymphoma; Refractory Angioimmunoblastic T-Cell Lymphoma; Refractory Mycosis Fungoides; Refractory Peripheral T-Cell Lymphoma, Not Otherwise Specified; Refractory Plasma Cell Myeloma; Refractory Primary Cutaneous T-Cell Non-Hodgkin Lymphoma; Refractory T-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Mycosis Fungoides; Multiple Myeloma; Lymphoma, T-Cell, Cutaneous; Lymphoma, T-Cell | interventions — Biopsy; Specimen Handling; Cyclophosphamide; Magnetic Resonance Spectroscopy; sodium-iodide symporter; X-Rays; Photons; cemiplimab; Immunoglobulin G; Disulfides; ruxolitinib; Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Group A (VSV-hIFNbeta-NIS, ruxolitinib) (Experimental): ** Group A no longer enrolling **
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Biological: Recombinant Vesicular Stomatitis Virus-expressing Human Interferon Beta and Sodium-Iodide Symporter; Procedure: Single Photon Emission Computed Tomography; Drug: Ruxolitinib; Procedure: Bone Marrow Aspiration
- Group B (VSV-hIFNbeta-NIS, ruxolitinib) (Experimental): ** Group B no longer enrolling **
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Biological: Recombinant Vesicular Stomatitis Virus-expressing Human Interferon Beta and Sodium-Iodide Symporter; Procedure: Single Photon Emission Computed Tomography; Drug: Ruxolitinib; Procedure: Multigated Acquisition Scan; Procedure: Echocardiography Test; Procedure: Bone Marrow Aspiration
- Group C (VSV-hIFNbeta-NIS, ruxolitinib, cyclophosphamide) (Experimental): ** Group C no longer enrolling **
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Procedure: Positron Emission Tomography; Biological: Recombinant Vesicular Stomatitis Virus-expressing Human Interferon Beta and Sodium-Iodide Symporter; Procedure: Single Photon Emission Computed Tomography; Drug: Ruxolitinib; Procedure: Bone Marrow Aspiration
- Group D (VSV-IFNbeta-NIS, rruxolitinib, nivolumab, ipilimumab) - MM only (Experimental): ** Group D no longer enrolling **
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Biological: Recombinant Vesicular Stomatitis Virus-expressing Human Interferon Beta and Sodium-Iodide Symporter; Procedure: Single Photon Emission Computed Tomography; Drug: Ruxolitinib; Biological: ipilimumab; Biological: Nivolumab; Procedure: Bone Marrow Aspiration
- Group E (VSV-IFNbeta-NIS, ruxolitinib, cemiplimab, ipilimumab - PTCL only (Experimental): PTCL patients receive cemiplimab IV over 30 minutes on day -3, ipilimumab IV over 30 minutes on day -3, VSV-hIFNβ-NIS IV over 30-60 minutes on day 1, and ruxolitinib PO on days 2-6 in the absence of disease progression or unacceptable toxicity. Patients also undergo PET/CT at baseline and then as clinically indicated, biopsy, and blood, buccal cell, and urine sample collection throughout the study. Patients undergo echocardiography or MUGA scan during screening as well as optional biopsy of imaging positive area on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Biological: Recombinant Vesicular Stomatitis Virus-expressing Human Interferon Beta and Sodium-Iodide Symporter; Procedure: Single Photon Emission Computed Tomography; Biological: Cemiplimab; Drug: Ruxolitinib; Biological: ipilimumab; Procedure: Multigated Acquisition Scan; Procedure: Echocardiography Test; Procedure: Bone Marrow Aspiration
- Group F (VSV-IFNbeta-NIS, ruxolitinib) - BCL Expansion Cohort (Experimental): BCL patients receive VSV-IFNbeta-NIS IV over 30 minutes on day 1 and ruxolitinib PO on days 2-6 in the absence of disease progression or unacceptable toxicity. Patients also undergo PET/CT during screening and as clinically indicated thereafter, bone marrow aspiration and biopsy, tumor or lymph node biopsy, and collection of blood, buccal cells, and urine throughout the study. Patients undergo echocardiography or MUGA scan during screening as well as optional biopsy of imaging positive area on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Biological: Recombinant Vesicular Stomatitis Virus-expressing Human Interferon Beta and Sodium-Iodide Symporter; Procedure: Single Photon Emission Computed Tomography; Drug: Ruxolitinib; Procedure: Multigated Acquisition Scan; Procedure: Echocardiography Test; Procedure: Bone Marrow Aspiration
- Group G (VSV-IFNbeta-NIS, ruxolitinib) - PTCL Expansion Cohort (Experimental): PTCL patients receive VSV-IFNbeta-NIS IV over 30 minutes on day 1 and ruxolitinib PO on days 2-6 in the absence of disease progression or unacceptable toxicity. Patients also undergo PET/CT during screening and as clinically indicated thereafter, bone marrow aspiration and biopsy, tumor or lymph node biopsy, and collection of blood, buccal cells, and urine throughout the study. Patients undergo echocardiography or MUGA scan during screening as well as optional biopsy of imaging positive area on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Biological: Recombinant Vesicular Stomatitis Virus-expressing Human Interferon Beta and Sodium-Iodide Symporter; Procedure: Single Photon Emission Computed Tomography; Drug: Ruxolitinib; Procedure: Multigated Acquisition Scan; Procedure: Echocardiography Test; Procedure: Bone Marrow Aspiration

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor or lymph node biopsy
  Other Names: Biopsy; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo SPECT/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
  Arms: Group C (VSV-hIFNbeta-NIS, ruxolitinib, cyclophosphamide)
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Biological: Recombinant Vesicular Stomatitis Virus-expressing Human Interferon Beta and Sodium-Iodide Symporter — Given IV
  Other Names: Oncolytic VSV-hIFNbeta-NIS; Vesicular Stomatitis Virus-expressing Human Interferon Beta and Sodium-Iodide Symporter; Voyager-V1; VSV-expressing hIFNb and NIS; VSV-hIFNb-NIS; VSV-hIFNbeta-NIS; VV1
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT/CT
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; Single-Photon Emission Computed; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; ST; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon
Biological: Cemiplimab — Given IV
  Other Names: 1801342-60-8; Cemiplimab RWLC; Cemiplimab-rwlc; Immunoglobulin G4; Anti-(Human Programmed Cell Death Protein 1) (Human Monoclonal REGN2810 Heavy Chain); Disulfide with Human Monoclonal REGN2810 kappa-chain; Libtayo; REGN2810; REGN-2810; REGN 2810
  Arms: Group E (VSV-IFNbeta-NIS, ruxolitinib, cemiplimab, ipilimumab - PTCL only
Drug: Ruxolitinib — Given PO
  Other Names: (3R)-3-cyclopentyl-3-(4-(7h-pyrrolo(2,3-d)pyrimidin-4-yl)pyrazol-1-yl)propanenitrile; 941678-49-5; INCB 018424; INCB-018424; INCB-18424; INCB18424; Oral JAK Inhibitor INCB18424
Biological: ipilimumab — Given IV
  Other Names: 477202-00-9; Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
  Arms: Group D (VSV-IFNbeta-NIS, rruxolitinib, nivolumab, ipilimumab) - MM only; Group E (VSV-IFNbeta-NIS, ruxolitinib, cemiplimab, ipilimumab - PTCL only
Biological: Nivolumab — Given IV
  Other Names: 946414-94-4; ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; ONO 4538; ONO-4538; ONO4538; Opdivo
  Arms: Group D (VSV-IFNbeta-NIS, rruxolitinib, nivolumab, ipilimumab) - MM only
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan, Equilibrium; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
  Arms: Group B (VSV-hIFNbeta-NIS, ruxolitinib); Group E (VSV-IFNbeta-NIS, ruxolitinib, cemiplimab, ipilimumab - PTCL only; Group F (VSV-IFNbeta-NIS, ruxolitinib) - BCL Expansion Cohort; Group G (VSV-IFNbeta-NIS, ruxolitinib) - PTCL Expansion Cohort
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC; Echocardiography
  Arms: Group B (VSV-hIFNbeta-NIS, ruxolitinib); Group E (VSV-IFNbeta-NIS, ruxolitinib, cemiplimab, ipilimumab - PTCL only; Group F (VSV-IFNbeta-NIS, ruxolitinib) - BCL Expansion Cohort; Group G (VSV-IFNbeta-NIS, ruxolitinib) - PTCL Expansion Cohort
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
  Other Names: bone marrow aspiratio

SUMMARY:
This phase I trial studies the best dose and side effects of the VSV-hIFNβ-NIS vaccine with or without cyclophosphamide and combinations of ipilimumab, nivolumab, and cemiplimab in treating patients with multiple myeloma, acute myeloid leukemia or lymphoma that has come back after a period of improvement (relapsed) or that does not respond to treatment (refractory). VSV-IFNβ-NIS is a modified version of the vesicular stomatitis virus (also called VSV). This virus can cause infection and when it does it typically infects pigs, cattle, or horses but not humans. The VSV used in this study has been altered by having two extra genes (pieces of DNA) added. The first gene makes a protein called NIS that is inserted into the VSV. NIS is normally found in the thyroid gland (a small gland in the neck) and helps the body concentrate iodine. Having this additional gene will make it possible to track where the virus goes in the body (which organs). The second addition is a gene for human interferon beta (β) or hIFNβ. Interferon is a natural anti-viral protein, intended to protect normal healthy cells from becoming infected with the virus. VSV is very sensitive to the effect of interferon. Many tumor cells have lost the capacity to either produce or respond to interferon. Thus, interferon production by tumor cells infected with VSV-IFNβ-NIS will protect normal cells but not the tumor cells. The VSV with these two extra pieces is referred to as VSV-IFNβ-NIS. Cyclophosphamide is in a class of medications called alkylating agents. It works by damaging the cell's DNA and may kill cancer cells. It may also lower the body's immune response. Immunotherapy with monoclonal antibodies, such as ipilimumab, nivolumab, and cemiplimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving VSV-IFNβ-NIS with or without cyclophosphamide and combinations of ipilimumab, nivolumab, and cemiplimab may be safe and effective in treating patients with recurrent peripheral T-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose (MTD) of recombinant vesicular stomatitis virus-expressing human interferon beta and sodium-iodide symporter (VSV-hIFNβ-NIS) in different treatment regimens (alone [Group A, F, G] in combination with ruxolitinib [Group B] and in combination with cyclophosphamide [Group C]) in patients with relapsed/refractory multiple myeloma, acute myeloid leukemia, T and B-cell lymphoma, or histiocytic/dendritic cell neoplasms; in combination with ipilimumab and nivolumab in patients with multiple myeloma [Group D] and in combination with ipilimumab and cemiplimab in patients with T-cell lymphoma [Group E].

SECONDARY OBJECTIVES:

I. To determine the safety profile of VSV-hIFNβ-NIS (alone and in combination). II. To estimate clinical response rate of VSV-hIFNβ-NIS (alone and in combination) in patients with relapsed/refractory multiple myeloma, acute myeloid leukemia, T and B-cell lymphoma, or histiocytic/dendritic cell neoplasms overall and by disease type.

III. To estimate progression-free and overall survival of VSV-hIFNβ-NIS (alone and in combination) in patients with relapsed/refractory multiple myeloma, acute myeloid leukemia, T and B-cell lymphoma, or histiocytic/dendritic cell neoplasms overall and by disease type.

CORRELATIVE OBJECTIVES:

I. To determine the time course of viral gene expression and virus elimination, and the biodistribution of virally infected cells at various times points after infection with VSV-hIFNβ-NIS using planar and single photon emission computed tomography (SPECT)/computed tomography (CT) or fluorine F 18 tetrafluoroborate (TFB)-positron emission tomography (PET) imaging.

II. To assess virus replication, viremia, viral shedding in urine and respiratory secretions, and virus persistence after systemic administration of VSV-hIFNβ-NIS.

III. To characterize the pharmacodynamics (PD) of VSV-IFNβ-NIS by way of measuring serum interferon-β and also vesicular stomatitis virus (VSV)-real time (RT)-polymerase chain reaction (PCR) of VSV-IFNβ-NIS.

IV. Assess CD8+ T cell (both general and VSV-IFNβ-NIS specific) and natural killer (NK) cell responses.

V. Gene expression analysis pre- and post-virotherapy. VI. Assess presence of VSV in tumor and normal tissues subsequent to administration of intravenous (IV) VSV-IFNβ-NIS.

VII. To identify the best dose of VSV-hIFNβ-NIS in the regimen being evaluated based on activity observed in the correlative measures described above in those dose levels identified as tolerable.

OUTLINE: This is a dose escalation study of VSV-hIFNβ-NIS followed by a dose-expansion study. Patients are assigned to 1 of 7 groups.

GROUP A: (CLOSED 7/30/2025)Patients receive VSV-hIFNβ-NIS IV over 30 minutes on day 1 and ruxolitinib PO on days 2-6 in the absence of disease progression or unacceptable toxicity. Patients also undergo PET/CT during screening and as clinically indicated thereafter, bone marrow aspiration and biopsy, tumor or lymph node biopsy, and collection of blood, buccal cells, and urine throughout the study. Patients may also receive optional TFB IV and undergo optional PET scan, as well as optional biopsy of imaging positive area on study.

GROUP B: Patients receive ruxolitinib PO on days -1 to 9 and VSV-hIFNβ-NIS IV over 30 minutes on day 1 in the absence of disease progression or unacceptable toxicity. Patients also undergo PET/CT during screening and as clinically indicated thereafter, bone marrow aspiration and biopsy, tumor or lymph node biopsy, and collection of blood, buccal cells, and urine throughout the study. Patients undergo echocardiography or multigated acquisition (MUGA) scan during screening as well as optional biopsy of imaging positive area on study.

GROUP C (CLOSED 7/30/2025): Patients receive ruxolitinib PO on days -1 to 9, VSV-hIFNβ-NIS IV over 30 minutes on day 1, and cyclophosphamide IV over 2 hours on day 2 in the absence of disease progression or unacceptable toxicity. Patients also undergo PET/CT during screening and as clinically indicated thereafter, bone marrow aspiration and biopsy, tumor or lymph node biopsy, and collection of blood, buccal cells, and urine throughout the study. Patients may also receive optional TFB IV and undergo optional PET scan, as well as optional biopsy of imaging positive area on study.

GROUP D (CLOSED 7/30/2025): Patients receive nivolumab IV over 30 minutes on day -3, ipilimumab IV over 30 minutes on day -3, VSV-hIFNβ-NIS IV over 30 minutes on day 1, and ruxolitinib PO on days 2-6 in the absence of disease progression or unacceptable toxicity. Patients also undergo PET/CT during screening and as clinically indicated thereafter, bone marrow aspiration and biopsy, tumor or lymph node biopsy, and collection of blood, buccal cells, and urine throughout the study. Patients may also receive optional TFB IV and undergo optional PET scan, as well as optional biopsy of imaging positive area on study.

GROUP E: Patients receive cemiplimab IV over 30 minutes on day -3, ipilimumab IV over 30 minutes on day -3, VSV-hIFNβ-NIS IV over 30-60 minutes on day 1, and ruxolitinib PO on days 2-6 in the absence of disease progression or unacceptable toxicity. Patients also undergo PET/CT at baseline and then as clinically indicated, biopsy, and blood, buccal cell, and urine sample collection throughout the study. Patients undergo echocardiography or MUGA scan during screening as well as optional biopsy of imaging positive area on study.

GROUP F: Patients receive VSV-hIFNβ-NIS IV over 30 minutes on day 1 and ruxolitinib PO on days 2-6 in the absence of disease progression or unacceptable toxicity. Patients also undergo PET/CT during screening and as clinically indicated thereafter, bone marrow aspiration and biopsy, tumor or lymph node biopsy, and collection of blood, buccal cells, and urine throughout the study. Patients undergo echocardiography or MUGA scan during screening as well as optional biopsy of imaging positive area on study.

GROUP G: Patients receive VSV-hIFNβ-NIS IV over 30 minutes on day 1 and ruxolitinib PO on days 2-6 in the absence of disease progression or unacceptable toxicity. Patients also undergo PET/CT during screening and as clinically indicated thereafter, bone marrow aspiration and biopsy, tumor or lymph node biopsy, and collection of blood, buccal cells, and urine throughout the study. Patients undergo echocardiography or MUGA scan during screening as well as optional biopsy of imaging positive area on study.

After completion of VSV-hIFNβ-NIS, patients are followed up on days 15 and 29, at 6 weeks, and then every 3 months until 1 year or until disease progression, whichever is longer, followed by every 6 months until a total of 2 years after registration.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Relapsed or refractory disease as follows:

  * Groups A, B, C or D: Multiple myeloma (MM) previously treated with an immunomodulatory imide drug (IMID), a proteosome inhibitor, and an alkylating agent
  * All Groups except D: Relapsed peripheral T-cell lymphoma (PTCL) of the following histologies: peripheral T-cell lymphoma-NOS (PTCL-NOS); angioimmunoblastic T-cell lymphoma (AITL), anaplastic large cell (ALCL), and mycosis fungoides (MF). Patients should have failed standard therapy and in the case of PTCL-NOS, AITL, and ALCL either have failed or be ineligible for high-dose therapy with autologous stem cell transplant
  * Group B and C only: B-cell lymphoma (other than Burkitt's lymphoma), or histiocytic/dendritic cell neoplasms (HCN) at any stage
  * Group E only: Relapsed peripheral T-cell lymphoma (PTCL) of the following histologies: peripheral T-cell lymphoma-NOS (PTCL-NOS); anaplastic large cell (ALCL), and mycosis fungoides (MF)
  * Group F only: Expansion Cohort for B-cell lymphoma (other than Burkitt's lymphoma) with low tumor burden
  * Group G only: Expansion Cohort for peripheral T cell lymphoma (PTCL) with low tumor burden
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2 times upper limit of normal (ULN) (obtained =< 15 days prior to registration)
* Creatinine =< 2.0 mg/dL (obtained =< 15 days prior to registration)
* Direct bilirubin =< 1.5 x ULN (obtained =< 15 days prior to registration)
* International normalized ratio (INR)/prothrombin time (PT) and activated partial thromboplastin time (aPTT) =< 1.5 x ULN (obtained =< 15 days prior to registration)
* If baseline liver disease, Child Pugh score not exceeding class A (obtained =< 15 days prior to registration)
* Negative pregnancy test for persons of child-bearing potential (obtained =< 15 days prior to registration)
* FOR MULTIPLE MYELOMA ONLY: Measurable disease of multiple myeloma as defined by at least ONE of the following:

  * Serum monoclonal protein >= 1.0 g/dL by protein electrophoresis
  * >= 200 mg of monoclonal protein in the urine on 24-hour electrophoresis
  * Serum immunoglobulin free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
* FOR MULTIPLE MYELOMA ONLY: Absolute neutrophil count (ANC) >= 1000/uL (obtained =< 14 days prior to registration)
* FOR MULTIPLE MYELOMA ONLY: Platelet (PLT) >= 100,000/uL (obtained =< 14 days prior to registration)
* FOR MULTIPLE MYELOMA ONLY: Hemoglobin >= 8.5 g/dl (obtained =< 14 days prior to registration)
* FOR AML ONLY: No ANC restriction (obtained =< 14 days prior to registration)
* FOR AML ONLY: PLT >= 10,000/uL (transfusion to get platelets >= 10,000 is allowed) (obtained =< 14 days prior to registration)
* FOR AML ONLY: Hemoglobin >= 7.5 g/dl (obtained =< 14 days prior to registration)
* FOR AML ONLY: Absence of uncompensated disseminated intravascular coagulation (DIC- as diagnosed by standard International Society on Thrombosis and Hemostasis [ISTH] criteria)
* FOR TCL/BCL ONLY: ANC >= 1,000/uL (obtained =< 14 days prior to registration)
* FOR TCL/BCL ONLY: PLT >= 100,000/uL (obtained =< 14 days prior to registration)
* FOR TCL/BCL ONLY: Hemoglobin >= 8.5 g/dl (obtained =< 14 days prior to registration)
* FOR TCL/BCL ONLY: Measurable disease by CT or magnetic resonance imaging (MRI): must have at least one lesion that has a single diameter of > 2 cm or tumor cells in the blood > 5 x 10^9/L; NOTE: skin lesions can be used if the area is > 2 cm in at least one diameter and photographed with a ruler and the images are available in the medical record
* FOR HCN ONLY: ANC >= 1,000/uL obtained =< 15 days prior to registration
* FOR HCN ONLY: PLT >= 100,000/uL obtained =< 15 days prior to registration
* FOR HCN ONLY: Hemoglobin >= 8.0 g/dl obtained =< 15 days prior to registration
* FOR HCN ONLY: Measurable disease by CT or MRI: Must have at least one lesion that has a single diameter of >= 1.5 cm or tumor cells in the blood >5 x10^9/L. NOTE: Skin lesions can be used if the area is >= 1.5 cm in at least one diameter and photographed with a ruler and the images are available in the medical record
* Absence of active central nervous system (CNS) involvement; NOTE: pre-enrollment lumbar puncture not mandatory
* Ability to provide written informed consent
* Willingness to return to Mayo Clinic for follow-up
* Life expectancy >= 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Willing to provide mandatory biological specimens for research purposes

Exclusion Criteria:

* Availability of and patient acceptance of curative therapy
* Uncontrolled infection
* Active tuberculosis or hepatitis, or chronic hepatitis
* Any of the following prior therapies:

  * Chemotherapy (IMIDs, alkylating agents, proteosome inhibitors) =< 2 weeks prior to registration
  * Immunotherapy (monoclonal antibodies) =< 4 weeks prior to registration
  * Experimental agent in case of AML or TCL within 4 half-lives of the last dose of the agent
* New York Heart Association classification III or IV, known symptomatic coronary artery disease, or symptoms of coronary artery disease on systems review, or known cardiac arrhythmias (atrial fibrillation or supraventricular tachycardia [SVT])
* Active CNS disorder or seizure disorder or known CNS disease or neurologic symptomatology; in case of AML active CNS involvement as detected by lumbar puncture or neuro-imaging (only to be done if clinically indicated)
* Human immunodeficiency virus (HIV) positive test result or other immunodeficiency or immunosuppression
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (used for a non-Food and Drug Administration [FDA] approved indication and in the context of a research investigation);

  * NOTE: in AML, the concurrent use of hydroxyurea to help control proliferative counts is allowed throughout the treatment protocol;
  * NOTE: in TCL, patients may use topical emollients or corticosteroids, acetic acid soaks, etc. to control pruritis and prevent infection; no topical chemotherapy is allowed (no topical nitrogen mustard)
* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women or women of reproductive ability who are unwilling to use effective contraception
  * Nursing women
  * Men who are unwilling to use a condom (even if they have undergone a prior vasectomy) while having intercourse with any woman, while taking the drug and for 4 weeks after stopping treatment
* AML ONLY: Current disseminated intravascular coagulopathy (DIC)
* ADDITIONAL EXCLUSION CRITERIA FOR GROUP A (LOW TUMOR BURDEN) ONLY:

  * Diagnosis of AML
  * Multiple myeloma only: > 25% plasma cells or plasmacytoma > 5cm in largest diameter
  * Lymphoma or HCN only: Any mass >5cm
  * Diagnosis of Burkitt's lymphoma
* ADDITIONAL EXCLUSION CRITERIA FOR GROUP B (HIGH TUMOR BURDEN) ONLY:

  * Diagnosis of AML
  * Diagnosis of Burkitt's lymphoma
* ADDITIONAL EXCLUSION CRITERIA FOR GROUP C (COMBINATION WITH CYCLOPHOSPHAMIDE) ONLY:

  * Diagnosis of AML
  * Diagnosis of Burkitt's lymphoma
* ADDITIONAL EXCLUSION CRITERIA FOR GROUP D AND E (COMBINATION WITH IPILIMUMAB AND NIVOLUMAB OR CEMIPLIMAB) ONLY:

  * Diagnosis of AML
  * Diagnosis of AITL
  * Hypersensitivity to ipilimumab or its excipients
* ADDITIONAL EXCLUSION CRITERIA FOR GROUP F (BCL EXPANSION COHORT) ONLY:

  * Diagnosis of Burkitt's lymphoma
* ADDITIONAL EXCLUSION CRITERIA FOR GROUP G (PTCL EXPANSION COHORT) ONLY:

  * Diagnosis of cutaneous TCL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Estimated)
Dates: Start 2017-04-04 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2032-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events of grade 3 or higher | Up to 2 years
  Assessed by the Common Terminology Criteria for Adverse Events version 4.0. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns (by cohort and overall). Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration. The rate of grade 3 or higher non-hematologic adverse events, and the rate of grade 4 or higher adverse event (hematologic and non-hematologic) will be computed each with a 95% exact binomial confidence.

SECONDARY OUTCOMES:
Clinical response | Up to 2 years
  The number of responses (complete response [CR], very good partial response, partial response [PR], or minimal response for multiple myeloma; CR, CR with incomplete recovery, cytogenetic complete response, PR for acute myeloid leukemia [AML]; CR or PR for T-cell lymphoma [TCL]) will be summarized by simple descriptive summary statistics.
Progression-free survival | From registration to disease progression or death due to any cause, assessed up to 2 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier (overall, by dose level, and by disease type).
Overall survival | From registration to death due to any cause, assessed up to 2 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier (overall, by dose level, and by disease type).

OTHER OUTCOMES:
Biodistribution and kinetics of virus spread | Up to 2 years
  Assessed by single photon emission computed tomography (SPECT)/computed tomography (CT) imaging. Descriptive statistics and scatterplots will form the basis of presentation of these variables. Correlations between the laboratory values and other outcome measures will be carried out by standard parametric and non-parametric tests (e.g., Pearson's and Spearman's rho). Will be correlated with tumor distribution.
NIS gene expression in tumor samples | Up to 2 years
  Assessed by single photon emission computed tomography (SPECT)/computed tomography (CT) imaging. Descriptive statistics and scatterplots will form the basis of presentation of these variables. Correlations between the laboratory values and other outcome measures will be carried out by standard parametric and non-parametric tests (e.g., Pearson's and Spearman's rho). Will be correlated with tumor distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Nora Bennani, M.D., Principal Investigator — Mayo Clinic in Rochester; Joselle Cook, M.B.B.S., Principal Investigator — Mayo Clinic in Rochester
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- [Result] Cook J, Peng KW, Witzig TE, Broski SM, Villasboas JC, Paludo J, Patnaik M, Rajkumar V, Dispenzieri A, Leung N, Buadi F, Bennani N, Ansell SM, Zhang L, Packiriswamy N, Balakrishnan B, Brunton B, Giers M, Ginos B, Dueck AC, Geyer S, Gertz MA, Warsame R, Go RS, Hayman SR, Dingli D, Kumar S, Bergsagel L, Munoz JL, Gonsalves W, Kourelis T, Muchtar E, Kapoor P, Kyle RA, Lin Y, Siddiqui M, Fonder A, Hobbs M, Hwa L, Naik S, Russell SJ, Lacy MQ. Clinical activity of single-dose systemic oncolytic VSV virotherapy in patients with relapsed refractory T-cell lymphoma. Blood Adv. 2022 Jun 14;6(11):3268-3279. doi: 10.1182/bloodadvances.2021006631. PMID 35175355
- [Derived] Macapagal SC, Bennani NN. Nodal peripheral T-cell lymphoma: Chemotherapy-free management, are we there yet? Blood Rev. 2023 Jul;60:101071. doi: 10.1016/j.blre.2023.101071. Epub 2023 Mar 3. PMID 36898933
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials